CLINICAL TRIAL: NCT00248430
Title: A Phase I-II Trial of Adoptive Immunotherapy Using Haploidentical, Related Donor-Lymphocyte Infusions and IL-2 After Autologous Stem Cell Transplantation for Advanced Lymphoid Malignancies
Brief Title: Donor White Blood Cell Infusions and Interleukin-2 in Treating Patients Who Are Undergoing an Autologous Stem Cell Transplant for Relapsed Advanced Lymphoid Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 1838.00; FHCRC-1838.00; CDR0000430694 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: graft versus host disease; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular | interventions — aldesleukin; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic allogeneic lymphocytes
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. An autologous stem cell transplant using the patient's stem cells may be able to replace blood-forming cells that were destroyed by chemotherapy. Giving white blood cells from a donor may help the patient's body destroy any remaining cancer cells. Interleukin-2 may stimulate the white blood cells to kill cancer cells.

PURPOSE: This phase I/II trial is studying the side effects of donor white blood cell infusions and interleukin-2 and to see how well they work in treating patients who are undergoing an autologous stem cell transplant for relapsed advanced lymphoid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and toxicity of haploidentical related donor lymphocyte infusions (DLI) and interleukin-2, in terms of acute graft-versus-host-disease, graft failure, and transplant-related mortality, in patients with relapsed advanced lymphoid malignancies undergoing autologous stem cell transplantation.

Secondary

* Determine the extent, degree, and duration of donor chimerism in patients treated with this regimen.
* Determine, preliminarily, activity of haploidentical DLI, as measured by complete response rate, in these patients.

OUTLINE: This is a pilot study.

Patients receive high-dose melphalan IV over 15-60 minutes on day -2 and undergo autologous stem cell transplantation on day 0. Patients receive haploidentical related donor lymphocyte infusions (DLI) IV on days 1, 5*, and 10* and interleukin-2 (IL-2) IV continuously on days 1-12.

NOTE: *DLI are not administered on days 5 or 10 if grade 3 or 4 graft-versus-host disease is present

After completion of study treatment, patients are followed monthly for 3 months and then every 3-12 months thereafter.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following advanced lymphoid malignancies:

  * Multiple myeloma, meeting both of the following criteria:

    * Deletion of chromosome 13
    * Elevated pre-transplant lactic dehydrogenase
  * Chronic lymphocytic leukemia (CLL)

    * Failed ≥ 2 prior conventional chemotherapy regimens, including fludarabine
  * Small lymphocytic lymphoma
  * Follicular non-Hodgkin's lymphoma

    * Received ≥ 3 prior conventional chemotherapy regimens
  * Mantle cell lymphoma

    * Received ≥ 3 prior conventional chemotherapy regimens
* Predicted poor outcome and relapsed disease after undergoing autologous stem cell transplantation ≥ 6 months ago
* Measurable disease, defined as any evidence of disease by scans or blood or urine analysis
* At least 8 x 10^6 autologous CD34-positive cells/kg available for transplantation

  * Stem cell mobilization allowed
* Haploidentical related donor available

  * Sex-mismatched
  * Identical for 1 HLA haplotype AND mismatched for ≥ 1 HLA-A, -B, -C, or DRB1 locus of the unshared haplotype
  * No HLA-identical related or unrelated donor available
* Not eligible for first-line autologous stem cell transplantation on protocol FHCRC-1368.00, FHCRC-1366.00, FHCRC-1461.00, or FHCRC-1595.00
* No bulky disease, defined as total volume of all measurable tumor > 500 cc
* No CNS disease resistant to therapy

PATIENT CHARACTERISTICS:

Age

* 18 to 69

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Liver function tests or liver enzymes ≤ 2 times upper limit of normal

Renal

* Not specified

Cardiovascular

* Ejection fraction ≥ 45%
* No symptomatic cardiac disease

Pulmonary

* DLCO ≥ 50%

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV Negative
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior allogeneic stem cell transplantation

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent contrast dye during and for 3 weeks after completion of interleukin-2 administration

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-08; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Feasibility
Toxicity

SECONDARY OUTCOMES:
Extent, degree, and duration of donor chimerism
Complete response rate

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington